CLINICAL TRIAL: NCT04701489
Title: Ultrasound Neural and Immunomodulation Treatment Evaluation Study (UMN-GE) for COVID-19
Brief Title: UNITE Study (UMN-GE) for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: General Electric Research (Industry); DARPA (Department of Defense) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: OTOL-2020-29216
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Covid19; Cytokine Storm; Inflammation
Keywords: ultrasound; ultrasound stimulation; spleen; immunomodulation; neuromodulation
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Inflammation

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to two groups: ultrasound group and control group. All participants will still receive standard clinical care. The ultrasound group will receive daily ultrasound application to the spleen for up to 7 days, in addition to the standard clinical care. The control group will receive standard clinical care without ultrasound stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Group (Experimental): Daily ultrasound application to the spleen of approximately 10 minutes for up to 7 days, in addition to standard clinical care.
  Interventions: Device: Splenic ultrasound
- Control Group (No Intervention): Standard clinical care with no ultrasound stimulation.

INTERVENTIONS:
Device: Splenic ultrasound — GE LOGIQ E10 device with C1-6 ultrasound probe
  Arms: Ultrasound Group

SUMMARY:
The research objective of the UNITE Study is to assess device feasibility of ultrasound application to the spleen to assess its effect on coronavirus disease 2019 (COVID-19) in a pilot study with an off-the-shelf ultrasound GE device originally used for diagnostic applications.

Specific Aims:

1. Determine the feasibility of splenic ultrasound with an ultrasound device in affecting physiological markers in COVID-19 infected patients between an ultrasound group versus a control group for the primary analyses; and
2. Evaluate the potential capabilities of splenic ultrasound in affecting additional outcomes in COVID-19 infected patients in the ultrasound group compared to a control group.

DETAILED DESCRIPTION:
Ultrasound is widely used in human medicine because it is safe, non-invasive, and painless. The same kind of ultrasound that is used for imaging (for example, to visualize babies in utero) may be able to treat inflammatory diseases including COVID-19. COVID-19 is a disease caused by infection with the SARS-CoV-2 virus. Some COVID-19 patients develop a severe respiratory disease called acute respiratory distress syndrome and this disease is caused, in part, by a significant increase in inflammatory factors. Clinical therapies that reduce this elevated inflammation in the body (e.g., inflammation molecules in your body called cytokines) may be capable of diminishing symptoms in severe cases of COVID-19.

Multiple studies in animals with hyper-inflammation conditions (e.g., inflammatory arthritis and sepsis/LPS injections) and recent human studies (e.g., for the treatment of joint inflammation in Rheumatoid Arthritis) have shown that ultrasound applied to the spleen can suppress blood/genetic markers of inflammation. Similar inflammatory markers, or cytokines, are elevated in the lungs of COVID-19 patients and believed to cause severe symptoms. Splenic ultrasound can potentially lower these inflammatory cytokines without hindering antibody production, leading to possible clinical improvements in COVID-19 patients.

This study will employ off-the-shelf ultrasound devices produced by General Electric (GE LOGIQ E10 device with C1-6 ultrasound probe) that are currently used in hospitals and approved for diagnostic imaging by the FDA. The ultrasound energies applied to the spleen in this study in COVID-19 patients will not exceed what is currently approved for diagnostic imaging with those GE ultrasound devices.

There will be two groups in this study with 15 participants in each group. One group will receive ultrasound application to the spleen, in addition to the standard clinical care. A control group will receive standard clinical care without splenic ultrasound. Each ultrasound application session will last about 15-20 minutes per day for 7 days, unless the participant is discharged sooner. For ultrasound stimulation, a small gel-coated probe is positioned on the upper left abdomen area over the ribs. The ultrasound session includes a period of 5-10 minutes when study personnel use the ultrasound device to locate the spleen and to position the ultrasound probe in a proper location around the ribs area, and an approximately 10-minute period for application of ultrasound to the spleen. Collection of various outcome data and daily blood draws will be performed in each participant throughout the study. Additional data collected from each participant during their routine clinical care beyond their study involvement will also be analyzed together with the study data to evaluate the specific aims of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Positive for SARS-CoV-2 (via PCR)
* Decreased blood oxygen saturation: Room air SaO2 < 94% and/or requiring supplemental oxygen to maintain SaO2 > 90%
* Admission to the hospital

Exclusion Criteria:

* Pregnant women
* Asplenia
* Ascites
* Open wound/sores near the stimulation site
* Recent abdominal surgery
* Splenomegaly
* Mechanically ventilated (if patient goes onto mechanical ventilation while participating in the study, they can continue ultrasound treatment if recommended by standard of care clinician and investigators of the study)
* Comfort care status
* Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
IL-6 changes | Baseline to Day 8 (end of stimulation; or date of discharge)
  Percentage of participants with observed change in IL-6 level
IL-1β changes | Baseline to Day 8 (end of stimulation; or date of discharge)
  Percentage of participants with observed change in IL-1β level
CRP changes | Baseline to Day 8 (end of stimulation; or date of discharge)
  Percentage of participants with observed change in CRP level

SECONDARY OUTCOMES:
Change in time to recovery | Baseline to date of recovery, assessed up to 21 days
  Day of recovery is defined as the first day on which the subject satisfies this category from the ordinal scale: Hospitalized, no oxygen therapy

OTHER OUTCOMES:
Change in death rate | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
Change in rate of requiring mechanical ventilation | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
Change in duration of hypoxemia | Baseline to date of discharge or date of death, whichever came first, assessed up to 6 months
Change in D-dimer levels | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in serum cytokine concentration of TNF | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in serum cytokine concentration of IL-10 | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in serum cytokine concentration of IFN-gamma | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in serum cytokine concentration of IL-18 | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in serum cytokine concentration of IL2R-alpha | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in serum cytokine concentration of IL-4 | Baseline to Day 8 (end of stimulation; or date of discharge)
Change in RNAseq identified pro-inflammatory pathways | Baseline to Day 8 (end of stimulation; or date of discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Lim, PhD, Principal Investigator — University of Minnesota
Locations (1):
- M Health Fairview St. Joseph's Hospital, Saint Paul, Minnesota, United States

REFERENCES:
- See also: First-in-human demonstration of splenic ultrasound stimulation for non-invasively controlling inflammation — https://www.medrxiv.org/content/10.1101/2020.07.14.20153528v2

DOCUMENTS (1):
  • Informed Consent Form (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT04701489/ICF_000.pdf